CLINICAL TRIAL: NCT03645980
Title: A Phase I/II Multicenter, Open-label Study of DKN-01 to Investigate the Anti-tumor Activity and Safety of DKN-01 in Patients With Hepatocellular Carcinoma and WNT Signaling Alterations
Brief Title: DKN-01 Inhibition in Advanced Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Leap Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. J. U. Marquardt, Jun. Prof. Dr. J. U. Marquardt, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Dial-1; 2017-002468-41 (EudraCT Number); AIO-HEP-0318 (Other: Arbeitsgemeinschaft Internistische Onkologie in der Deutschen Krebsgesellschaft e.V (AIO))
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: DKN-01; Hepatocellular Carcinoma; WNT signaling
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKN-01 300 mg (Experimental): Phase I Study treatment will be started as monotherapy with DKN-01 for up to 8 weeks or until unacceptable toxicity occurs. The study will be continued as combination therapy of DKN-01 and sorafenib until objective disease progression (PD) or unacceptable toxicity occurs. The dose of DKN-01 for cohort 1 will be 300 mg , depending on the results of the safety assessment. Phase II The dose of DKN-01 will be the recommended phase II dose (RP2D) determined from Part A. Study treatment will be started as monotherapy with DKN-01 until objective disease progression (PD1) or unacceptable toxicity occurs. After PD1, study treatment will be continued as combination therapy of DKN-01 and sorafenib until disease progression (PD2) or unacceptable toxicity occurs.
  Interventions: Drug: DKN-01 300 mg; Drug: Sorafenib
- DKN-01 600 mg (Experimental): Phase I Study treatment will be started as monotherapy with DKN-01 for up to 8 weeks or until unacceptable toxicity occurs. The study will be continued as combination therapy of DKN-01 and sorafenib until objective disease progression (PD) or unacceptable toxicity occurs. The dose of DKN-01 for cohort 2 will be 600 mg or 150 mg, depending on the results of the safety assessment. Phase II The dose of DKN-01 will be the recommended phase II dose (RP2D) determined from Part A. Study treatment will be started as monotherapy with DKN-01 until objective disease progression (PD1) or unacceptable toxicity occurs. After PD1, study treatment will be continued as combination therapy of DKN-01 and sorafenib until disease progression (PD2) or unacceptable toxicity occurs.
  Interventions: Drug: DKN-01 600 mg; Drug: Sorafenib

INTERVENTIONS:
Drug: DKN-01 300 mg — DKN-01 will be administered intravenous (IV) over a minimum of 30 minutes and up to a maximum of 2 hours given on days 1 and 15 of each 28 day cycle.
  Arms: DKN-01 300 mg
Drug: DKN-01 600 mg — DKN-01 will be administered intravenous (IV) over a minimum of 30 minutes and up to a maximum of 2 hours given on days 1 and 15 of each 28 day cycle.
  Arms: DKN-01 600 mg
Drug: Sorafenib — For combination with DKN-01, sorafenib will be administrated according to standard clinical practice. Part A: After 8 weeks monotherapy with DKN-01, the study will be continued as combination therapy of DKN-01 and sorafenib until objective disease progression (PD) or unacceptable toxicity occurs. Part B:After PD1, study treatment will be continued as combination therapy of DKN-01 and sorafenib until disease progression (PD2) or unacceptable toxicity occurs.

SUMMARY:
This clinical trial is a prospective, open label, single arm oncological phase I/II trial in patients with hepatocellular carcinoma and WNT signaling alterations. The trial consists of two parts: Part A is a phase I study investigating the safety of DKN-01 administered as mono- as well as combination therapy with sorafenib in a 2 step dose escalation.Part B is a phase II study to investigate the anti-tumor activity and safety of DKN-01 in patients with advanced HCC. DKN-01 is administered at the recommend phase II dose (RP2D) for monotherapy and at the recommend phase II dose for combination therapy established in Part A.

DETAILED DESCRIPTION:
Part A is a phase I study investigating the safety of DKN-01 administered as mono- as well as combination therapy with sorafenib in a 2 step dose escalation. Up to 20 patients with advanced HCC will be included in Part A. Tumor assessment will be performed every 8 weeks.The first 10 patients (cohort 1) will start with IV infusion of 300 mg DKN-01 on day 1 and 15 (monotherapy for 28 days). DLTs will be determined. After cycle 2 of monotherapy patients of cohort 1 will continue with combination of 300 mg DKN-01 IV on day 1 and 15 and sorafenib (recommended dose 800 mg per day or at discretion of the investigator) until disease progression. After 2 cycles of combination therapy and prior to the start of the next cohort DLTs will be determined. Part B is a phase II study to investigate the anti-tumor activity and safety of DKN-01 in patients with advanced HCC. DKN-01 is administered at the recommend phase II dose (RP2D) for monotherapy and at the recommend phase II dose for combination therapy established in Part A. Depending on the tolerability, the doses may be different for monotherapy and for combination therapy. Up to 50 additional patients with advanced HCC may be enrolled in Part B. Every 8 weeks tumor assessment will be performed. If progression of disease (PD1) is observed with DKN-01 monotherapy, patients will continue on study receiving DKN-01 at the recommend phase II dose for combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female patients ≥ 18 years
* Patients must have histologically confirmed diagnosis (by either primary surgical specimen or biopsy for recurrence) of advanced stage or recurrent diagnosis of HCC based on histopathologic findings.
* Tumor tissue is mandatory for pre-treatment evaluation (baseline) (fresh biopsy during 4-weeks screening time preferred. Archived specimen is only acceptable, if ≤ 6 months old. Baseline tumor biopsy samples must be available prior to the first dose of DKN-01.
* Tumor tissue (FFPE) must be received by central histopathology laboratory for correlative studies (fine needle aspiration and bone metastasis samples are not acceptable).
* Patients with activated WNT/β-catenin signaling identified by glutamine synthetase staining (high positive staining in tumor tissue) by an approved lab. Positive staining must be confirmed prior to first dose of DKN-01.
* Child-Pugh score <7 (Child-Pugh Class A).
* Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to resection, locoregional therapy or refractory to locoregional therapy.
* At least one tumor lesion measurable on radiographic imaging as defined by mRECIST for HCC that has not been previously treated by locoregional therapies.
* Locoregional therapies or radiation therapy must be completed at least 4 weeks prior to baseline scan. All toxic effects > grade 1 (NCI CTCAE v5.0) related to any prior HCC treatment must be resolved. Palliative radiotherapy for symptomic control is acceptable and no additional radiotherapy for the same lesion is planned. (like bone metastases should not be targets for RECIST).
* ECOG performance status (PS) of 0 or 1.
* Estimated life expectancy of at least 3 months, in the judgment of the Investigator.
* Disease-free of active second/secondary or prior malignancies for ≥2 years with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast.
* Patients are eligible to enroll if they have non-viral-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

  * HBV-HCC: Resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Patients with chronic HBV infection must have HBV DNA < 2000 IU/mL and must be on antiviral therapy.
  * HCV-HCC: Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody
* Acceptable liver function:

  * Total bilirubin ≤2.0 × upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 × ULN.
* Acceptable renal function:

  o Calculated creatinine clearance ≥50 mL/min using the Cockcroft and Gault Method (Cockroft and Gault 1976).
* Acceptable hematologic status:

  * Neutrophil Granulocyte ≥1500 cells/μl.
  * Hemoglobin ≥ 8,5 g/dL (transfusion permitted within 30 days of study entry).
  * Platelet count ≥75,000 cells/μl.
* Acceptable coagulation status:

  o INR ≤ 1.7 and no active bleeding, (i.e., no clinically significant bleeding within 14 days prior to first dose of study therapy
* Female subjects who are post-menopausal (defined as spontaneous amenorrhea for at least a year) or permanently sterilized (e.g. bilateral oophorectomy, hysterectomy, bilateral salpingectomy) can participate in the trial and are not required to use any contraception.
* Women of child bearing potential (WOCBP, a woman is considered of childbearing potential i.e. fertile, following menarche and until becoming post-menopausal) must have a negative serum or urine pregnancy test within 7 days prior to first dose of DKN- 01. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG.
* Women of childbearing potential must be willing to practice a highly effective and medically accepted contraception method during trial and for 18 months after last dose of study drug. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as:

  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
  * progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system ( IUS)
  * bilateral tubal occlusion
  * vasectomised partner (medical assessment must be present and done)
  * sexual abstinence when this is in line with the preferred and usual lifestyle of the subject
* Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method (LAM) are not acceptable methods of contraception. Female condom and male condom should not be used together.
* Sexually-active male subjects must be willing to use contraception (condom, contraception for non-pregnant WOCBP partner) with their partners throughout the study and for 18 months after last dose of study drug and agree to inform the Investigator if the respective partner becomes pregnant during this time
* Provided written informed consent prior to any study-specific procedures.
* Ability of patient to understand nature, importance and individual consequences of clinical trial.

Exclusion Criteria:

* Patients with the following histology of hepatocellular cancer are not eligible for enrollment: fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma.
* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
* Specific cardiac preconditions : Fridericia-corrected QT interval (QTcF) >470 msec (female) or >450 msec (male), or history of congenital long QT syndrome. Any ECG abnormality that in the opinion of the Investigator would preclude safe participation in the study; patients with pacemakers where QTc is not a reliable measure will require an evaluation by a cardiologist to exclude co-existing cardiac conditions which would prohibit safe participation in the study.
* Active, uncontrolled bacterial, viral, or fungal infections, within 7 days of study entry requiring systemic therapy.
* Known to be human immunodeficiency virus (HIV) positive,
* History of major organ transplant (i.e., heart, lungs, liver, or kidney).
* History of autologous/allogenic bone marrow transplant.
* Serious non-malignant disease that could compromise protocol objectives in the opinion of the Investigator and/or Sponsor.
* Pregnancy or nursing.
* Major surgical procedures, open biopsy or significant traumatic injury within 4 weeks prior to treatment start (minor procedures within 1 week)
* History of osteonecrosis of the hip or evidence of structural bone abnormalities in the proximal femur on magnetic resonance imaging (MRI) scan that are symptomatic and clinically significant. Degenerative changes of the hip joint are not exclusionary. Screening of asymptomatic patients is not required.
* Symptomatic central nervous system (CNS) malignancy or metastasis. Patients with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic patients without a history of CNS metastases is not required.
* Known osteoblastic bone metastasis. Screening of asymptomatic patients without a history of metastatic bone lesions is not required.
* Medical or psychological conditions that would jeopardise an adequate and orderly completion of the trial.
* Thrombotic or embolic events (except HCC tumor thrombus <pVT4) within the past 6 months (including cerebrovascular accidents)
* Evidence of portal hypertension with bleeding esophageal or gastric varices within the past 6 months
* Patients with portal vein thrombosis = pVT4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Adverse Events | assessment period is 2 cycles for monotherapy (each cycle is 28 days)
  Absolute and relative incidences of treatment-emergent adverse events.
Phase I: Adverse Events | assessment period is 2 cycles for combination therapy (each cycle is 28 days)
  Absolute and relative incidences of treatment-emergent adverse events.
Phase II: Time to progression (TTP2) | time from the first DKN-01 intake until PD2, assessed up to 2 years
  The TTP2 is defined as the time from the first DKN-01 intake until PD2. Tumor progression is assessed by mRECIST criteria (modified Response Evaluation Criteria in Solid Tumors).

SECONDARY OUTCOMES:
Phase I: pharmacokinetics of DKN-01 | monotherapy for 8 weeks and in combination with sorafenib for 8 weeks
  Serum DKN-01 levels to characterize the pharmacokinetics of DKN-01 when administered at the dose of 300 mg and 600 mg as monotherapy and in combination with sorafenib
Phase II: Overall survival (OS) | time from first DKN-01 intake until death from any cause, assessed up to 2 years
  Overall survival is defined as the time from first DKN-01 intake until death from any cause, assessed up to 2 years
Phase II: progression free survival (PFS1, PFS2) | time from first DKN- 01 intake until death or PD1 or PD2 respectively whichever comes first, assessed up to 2 years
  Progression free survival (PFS1, PFS2) is defined as the time from first DKN-
  01 intake until death or PD1 or PD2 respectively whichever comes first, assessed up to 2 years
Phase II:objective response rate (ORR) | 2, 4 and 6 months after first DKN- 01 intake
  ORR (CR or PR), binary measurement
Phase II: disease control rate (DCR) | 2, 4 and 6 months after first DKN- 01 intake
  DCR (CR, PR or SD), binary measurement (CR, PR or SD) after 2, 4 and 6 months will be analyzed by absolute and relative frequencies.
Phase II: Duration of disease control with DKN-01 | time from first to the last disease control (CR, PR, or SD), assessed up to 2 years
  Duration of disease control is defined as the time from the first to the last occurrence of disease control (CR, PR, or SD), assessed up to 2 years
Phase II: Adverse Events | assessment period is during mono- and combination therapy with sorafenib (through study completion, estimated 2 years)
  Absolute and relative incidences of treatment-emergent adverse events as assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jens U Marquardt, Dr med, Principal Investigator — Universitätsklinikum Schleswig Holstein Campus Lübeck
Locations (6):
- Germany (6):
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Med. Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig Holstein Campus Lübeck, Lübeck
  - Universitätsmedizin Mainz, I. Med. Klinik und Poliklinik, Mainz
  - II. Medizinische Universitätsklinik Gastroenterologie, Hepatologie, Infektiologie, Mannheim